CLINICAL TRIAL: NCT06778720
Title: Implementing Music Therapy for Video-Assisted Thoracoscopic Surgery Patients: A Quality Improvement Initiative
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Sandra Nahom, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003902
Record Dates: First submitted 2025-01-09; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Pain Assessment; VATS; Music Therapy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music Therapy (Experimental): Participants receive music therapy as an evidence-based pain management practice to reduce pain levels in the PACU after a VATS procedure.
  Interventions: Behavioral: Music Therapy with over-the ear headphones

INTERVENTIONS:
Behavioral: Music Therapy with over-the ear headphones — Eligible patients undergoing VATS procedure can have music therapy as an intervention to reduce pain levels after surgery and improve outcomes.

SUMMARY:
The purpose of this project is to introduce and implement music therapy as an evidence-based pain management protocol focused on reducing postoperative pain levels among Video-Assisted Thoracoscopic Surgery (VATS) patients in the Post-Anesthesia Care Unit (PACU) of the project site. The clinical question guiding this initiative is: In adult patients undergoing a VATS procedure, does the implementation of music therapy lead to lower postoperative pain scores in the PACU compared to no intervention within an 8-week timeframe? The investigator will ask eligible patients their immediate pain scores upon arrival into the PACU and then start music of patient's choice via over-the-ear headphones. Pain scores will be rechecked 30 minutes after implementation of music therapy. The standard of care pain medications and/or usual care will not be withheld or altered after surgery in lieu of music therapy.

DETAILED DESCRIPTION:
The clinical question guiding this initiative is: In adult patients undergoing a VATS procedure, does the implementation of music therapy lead to lower postoperative pain scores in the PACU compared to no intervention within an 8-week timeframe? The investigator will ask eligible patients their immediate pain scores upon arrival into the PACU and then start music of patient's choice via over-the-ear headphones. Pain scores will be rechecked 30 minutes after implementation of music therapy. The standard of care pain medications and/or usual care will not be withheld or altered after surgery in lieu of music therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older with lung mass diagnosis undergoing VATS

Exclusion Criteria:

* Individuals with dementia, neurocognitive disorders, or chronic pain conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-14 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
Changes in pain scores after implementation, as measured by Numerical Rating Scale (NRS) | Principal investigator will introduce intervention in the preoperative area prior to surgery. Then participant will have scheduled VATS procedure. Then the assessment will take place immediately following the surgery in the PACU.
  Measuring pain scores of VATS patients immediately after arrival to PACU. After music therapy is implemented, pain scores will be repeated after 30 minutes to see if there is an improvement of pain due to music implementation. Pain will be measured using the Numerical Rating Scale (NRS) pain assessment tool.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Nahom, MSN, RN, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
I do not plan to publish results. This is for a school project.

REFERENCES:
- [Background] Zhang QL, Xu N, Huang ST, Lin ZW, Chen LW, Cao H, Chen Q. Music Therapy for Early Postoperative Pain, Anxiety, and Sleep in Patients after Mitral Valve Replacement. Thorac Cardiovasc Surg. 2020 Sep;68(6):498-502. doi: 10.1055/s-0040-1713352. Epub 2020 Jun 30. PMID 32604430
- [Background] Thaut MH. Music as therapy in early history. Prog Brain Res. 2015;217:143-58. doi: 10.1016/bs.pbr.2014.11.025. Epub 2015 Jan 31. PMID 25725914
- [Background] Patiyal N, Kalyani V, Mishra R, Kataria N, Sharma S, Parashar A, Kumari P. Effect of Music Therapy on Pain, Anxiety, and Use of Opioids Among Patients Underwent Orthopedic Surgery: A Systematic Review and Meta-Analysis. Cureus. 2021 Sep 29;13(9):e18377. doi: 10.7759/cureus.18377. eCollection 2021 Sep. PMID 34725621
- [Background] Lin CL, Hwang SL, Jiang P, Hsiung NH. Effect of Music Therapy on Pain After Orthopedic Surgery-A Systematic Review and Meta-Analysis. Pain Pract. 2020 Apr;20(4):422-436. doi: 10.1111/papr.12864. Epub 2020 Jan 9. PMID 31785131
- [Background] Liang J, Tian X, Yang W. Application of Music Therapy in General Surgical Treatment. Biomed Res Int. 2021 Sep 28;2021:6169183. doi: 10.1155/2021/6169183. eCollection 2021. PMID 34621896
- [Background] Li G, Yu L, Yang Y, Deng J, Shao L, Zeng C. Effects of Perioperative Music Therapy on Patients with Postoperative Pain and Anxiety: A Systematic Review and Meta-Analysis. J Integr Complement Med. 2024 Jan;30(1):37-46. doi: 10.1089/jicm.2022.0803. Epub 2023 Aug 30. PMID 37646752
- [Background] Laframboise-Otto JM, Horodyski M, Parvataneni HK, Horgas AL. A Randomized Controlled Trial of Music for Pain Relief after Arthroplasty Surgery. Pain Manag Nurs. 2021 Feb;22(1):86-93. doi: 10.1016/j.pmn.2020.09.003. Epub 2020 Oct 28. PMID 33129705
- [Background] Komann M, Weinmann C, Schwenkglenks M, Meissner W. Non-Pharmacological Methods and Post-Operative Pain Relief: An Observational Study. Anesth Pain Med. 2019 Apr 20;9(2):e84674. doi: 10.5812/aapm.84674. eCollection 2019 Apr. PMID 31341822
- [Background] Kahloul M, Mhamdi S, Nakhli MS, Sfeyhi AN, Azzaza M, Chaouch A, Naija W. Effects of music therapy under general anesthesia in patients undergoing abdominal surgery. Libyan J Med. 2017 Dec;12(1):1260886. doi: 10.1080/19932820.2017.1260886. PMID 28452603
- [Background] Dale VH. The impact of perioperative music on abdominal surgery patients' experience of postoperative pain: A systematic review and meta-analysis. J Perioper Pract. 2021 Jan-Feb;31(1-2):31-43. doi: 10.1177/1750458920943375. Epub 2020 Sep 8. PMID 32894995
- [Background] Choi EK, Baek J, Lee D, Kim DY. Effect on music therapy on quality of recovery and postoperative pain after gynecological laparoscopy. Medicine (Baltimore). 2023 Mar 3;102(9):e33071. doi: 10.1097/MD.0000000000033071. PMID 36862891
- [Background] Bojorquez GR, Jackson KE, Andrews AK. Music Therapy for Surgical Patients: Approach for Managing Pain and Anxiety. Crit Care Nurs Q. 2020 Jan/Mar;43(1):81-85. doi: 10.1097/CNQ.0000000000000294. PMID 31789881